CLINICAL TRIAL: NCT02974998
Title: Expanding HIV Testing and Prevention to Reach Vulnerable Young Women
Brief Title: Cape Town Young Women's Health CoOp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA041227 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Condomless Sex; Human Immunodeficiency Virus (HIV); Sexually Transmitted Infections (STIs); Alcohol and Drug Use; Violence and Victimization; Access and Linkage to Healthcare; Education Advancement
Keywords: Human Immunodeficiency Virus (HIV); HIV Testing and Counseling (HTC); Sexually Transmitted Infections (STIs); Substance Abuse; Gender Based Violence; Gang Violence; Victimization; Linkage to Care; Sexual Risk; Out-of-school Adolescents; Young Women
MeSH Terms: conditions — Unsafe Sex; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young Women's Health CoOp (YWHC)/ HTC (Experimental): Participants received an enhanced gender-focused HTC intervention.
  Interventions: Behavioral: Young Women's Health CoOp (YWHC)
- Standard HTC (Active Comparator): Participants received the standard HTC available in South Africa for this population.
  Interventions: Behavioral: Standard HTC

INTERVENTIONS:
Behavioral: Young Women's Health CoOp (YWHC) — Participants received HTC and engaged in a two-session gender-focused intervention. The intervention included information addressing the intersection of substance use, sexual risk, and violence through skill building, role-play, and rehearsal. The intervention also encouraged positive goal-seeking to access linkages to health care within the larger social ecological framework of where the young women live.
  Arms: Young Women's Health CoOp (YWHC)/ HTC
Behavioral: Standard HTC — Participants received the standard HTC available in South Africa for this population.
  Arms: Standard HTC

SUMMARY:
This two-arm cluster randomized trial tested a gender-focused comprehensive HIV testing and counselling (HTC) program, the Young Women's Health CoOp (YWHC) with a standard HTC program and targeted female adolescents (aged 16-19) who use substances and have dropped out of school. To evaluate the process, the study examined the feasibility of using peer role models as recruiters and co-facilitators of the intervention and monitored fidelity to the intervention. Efficacy of the intervention on behavioral and biological outcomes, and on linkages to health services, through follow-up visits conducted 6- and 12-months post-enrollment was also assessed.

DETAILED DESCRIPTION:
The purpose of this study was to test a gender-focused comprehensive HIV testing and counselling (HTC) program, the Young Women's Health CoOp (YWHC) with a standard HTC program in 24 disadvantaged communities in Cape Town, South Africa. The researchers conducted community-level randomization across the 24 communities with balanced recruitment from predominantly Black African and predominantly Coloured communities. The aims of the study were: Aim 1. To train and evaluate adolescent peer role models to conduct community outreach with established outreach workers to recruit 500 out-of-school, substance-using female adolescents aged 16 to 19 for HIV testing and counseling (HTC) and to co-facilitate a gender-focused comprehensive HTC program. Aim 2. To test the efficacy of a young women's gender-focused comprehensive HTC program for reducing substance use, victimization, and sexual risk behavior (primary outcomes) and improving access to effective treatment and support services through linkages to care (substance abuse treatment, HIV, sexually transmitted infections [STIs], antenatal and reproductive health as secondary outcomes) relative to standard HTC for adolescent females. The Young Women's Health CoOp has been adapted from the South African Women's Health CoOp (WHC) and the North Carolina Young Women's CoOp (YWC) which was found acceptable in focus groups and maintained all the core elements of the evidence-based intervention. For this study, the intervention was co-facilitated by trained staff from the local communities. The intervention consisted of two 1.5-hour group workshops (sessions), each having several modules that are usually administered a week apart: Workshop 1: Developmental Issues and Alcohol and Other Drugs; Gender, Problem-Solving and Conflict Negotiation, Violence and Values and Becoming a Powerful Young Woman: and Workshop 2: STIs, HIV/AIDS, Prevention, Condoms and Role-play. After each session, each participant developed a risk-reduction personalized action plan (PAP). To maintain PAP goals and reduce decay of intervention effects over time, the staff conducted case management to help participants attain these personal goals. Participants completed baseline, 6-month follow-up and 12-month follow-up assessments, which included a survey and biological testing for substance use, pregnancy and HIV.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Self-identify as living in one of the 24 targeted disadvantaged communities
* Between 16 and 19 years old
* Has dropped out of school for at least 6 months
* Is currently dropped out of school
* Has not completed matric (high school diploma) or have an N3 Certificate (South Africa National Technical Certificate)
* Reports consuming 2-3 alcoholic drinks at least once in the last 30 days or using illicit drugs at least once a week.
* Reports unprotected sex with a male partner in the last 90 days
* Is able to provide informed assent to participate or informed consent if emancipated or 18 years old
* Has lived in targeted community for at least 6 months and plans to reside in the target community for the next year and provide verifiable locator information

Exclusion Criteria:

* Participant must be able to pass a cognitive test

Ages: 16 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2016-11; Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Reduced Sexual Risk | Baseline
  Reduced drug or alcohol use prior to sex (impairment), self-reported number of casual partners, sex trading, and concurrent partners (defined ≥ 2 partners in past 90 days) measured by the PRBA (WHC Pretoria Risk Behavior Assessment)
Reduced Sexual Risk | 6 months after baseline
  Reduced drug or alcohol use prior to sex (impairment), self-reported number of casual partners, sex trading, and concurrent partners (defined ≥ 2 partners in past 90 days) measured by the PRBA (WHC Pretoria Risk Behavior Assessment
Reduced Sexual Risk | 12 months after baseline
  Reduced drug or alcohol use prior to sex (impairment), self-reported number of casual partners, sex trading, and concurrent partners (defined ≥ 2 partners in past 90 days) measured by the PRBA (WHC Pretoria Risk Behavior Assessment
Increased Condom Use | Baseline
  Reduced number of unprotected anal and vaginal sex acts in the past 90 days. Increased skillful condom communication as measured by the 3-item Condom Negotiation scale measured by the YRBA (Youth revised Risk Behavior Assessment)
Increased Condom Use | 6 months after baseline
  Reduced number of unprotected anal and vaginal sex acts in the past 90 days. Increased skillful condom communication as measured by the 3-item Condom Negotiation scale measured by the YRBA (Youth revised Risk Behavior Assessment)
Increased Condom Use | 12 months after baseline
  Reduced number of unprotected anal and vaginal sex acts in the past 90 days. Increased skillful condom communication as measured by the 3-item Condom Negotiation scale measured by the YRBA (Youth revised Risk Behavior Assessment)
Reduced Alcohol and Illicit Drug Use | Baseline
  Self-reported frequency of alcohol and illicit drug use the past 30 days as measured by PRBA. Biological measures of drug use through urine drug tests and breathalyzer tests.
Reduced Alcohol and Illicit Drug Use | 6 months after baseline
  Self-reported frequency of alcohol and illicit drug use the past 30 days as measured by PRBA. Biological measures of drug use through urine drug tests and breathalyzer tests.
Reduced Alcohol and Illicit Drug Use | 12 months after baseline
  Self-reported frequency of alcohol and illicit drug use the past 30 days as measured by PRBA. Biological measures of drug use through urine drug tests and breathalyzer tests.
Reduced Violence and Victimization | Baseline
  Self-reported recent emotional, physical, and sexual abuse in the past 6 months measured by the RRBA (WHC Revised Risk Behavior Assessment).
Reduced Violence and Victimization | 6 months after baseline
  Self-reported recent emotional, physical, and sexual abuse in the past 6 months measured by the RRBA (WHC Revised Risk Behavior Assessment).
Reduced Violence and Victimization | 12 months after baseline
  Self-reported recent emotional, physical, and sexual abuse in the past 6 months measured by the RRBA (WHC Revised Risk Behavior Assessment).

SECONDARY OUTCOMES:
Increased Access to Health Services | Baseline
  Self-reported use of sexual reproductive health and HIV & STI testing services; linkage to HIV treatment and care services, staging and antiretroviral therapy (ART) initiation.
Increased Access to Health Services | 6 months after baseline
  Self-reported use of sexual reproductive health and HIV & STI testing services; linkage to HIV treatment and care services, staging and antiretroviral therapy (ART) initiation.
Increased Access to Health Services | 12 months after baseline
  Self-reported use of sexual reproductive health and HIV & STI testing services; linkage to HIV treatment and care services, staging and antiretroviral therapy (ART) initiation.
Increased Advancement in Education and Job Training | Baseline
  Enrollment in training certifications; self-reported motivation and perception regarding learning; self-reported knowledge regarding strategies to improve educational outcomes.
Increased Advancement in Education and Job Training | 6 months after baseline
  Enrollment in training certifications; self-reported motivation and perception regarding learning; self-reported knowledge regarding strategies to improve educational outcomes.
Increased Advancement in Education and Job Training | 12 months after baseline
  Enrollment in training certifications; self-reported motivation and perception regarding learning; self-reported knowledge regarding strategies to improve educational outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (1):
- The South African Medical Research Council (SAMRC),, Cape Town, South Africa

REFERENCES:
- [Background] Wechsberg WM, Browne FA, Carney T, Myers B, Minnis A, MacDonald R, Ndirangu JW, Turner LB, Howard BN, Rodman N. The Young Women's Health CoOp in Cape Town, South Africa: Study protocol for a cluster-randomised trial for adolescent women at risk for HIV. BMC Public Health. 2018 Jul 11;18(1):859. doi: 10.1186/s12889-018-5665-5. PMID 29996792
- [Result] Bonner CP, Fisher CB, Carney T, Browne FA, Gichane MW, Howard BN, Turner L, Wechsberg WM. "Because all mothers is not the same": The development and implementation of an in loco parentis informed consent procedure to enroll adolescent girls and young women to participate in HIV research. J Adolesc. 2021 Dec;93:234-244. doi: 10.1016/j.adolescence.2021.11.001. Epub 2021 Dec 9. PMID 34896961
- [Result] Myers B, Browne FA, Carney T, Kline T, Bonner CP, Wechsberg WM. The Association of Recurrent and Multiple Types of Abuse with Adverse Mental Health, Substance Use, and Sexual Health Outcomes among Out-of-School Adolescent Girls and Young Women in Cape Town, South Africa. Int J Environ Res Public Health. 2021 Oct 29;18(21):11403. doi: 10.3390/ijerph182111403. PMID 34769920
- [Result] Bonner CP, Carney T, Browne FA, Ndirangu JW, Howard BN, Wechsberg WM. Substance use and depressive and anxiety symptoms among out-of-school adolescent girls and young women in Cape Town, South Africa. S Afr Med J. 2020 Dec 14;111(1):40-45. doi: 10.7196/SAMJ.2020.v111i1.14520. PMID 33404004
- [Result] Bonner CP, Browne FA, Carney T, Shangase N, Ndirangu JW, Myers B, Wechsberg WM. Mandrax use, sexual risk, and opportunities for pre-exposure prophylaxis among out-of-school adolescent girls and young women in Cape Town, South Africa. S Afr Med J. 2022 Apr 29;112(5):341-346. PMID 35587247
- [Derived] Wechsberg WM, Browne FA, Carney T, Kline TL, Howard BN, Russell SE, van der Drift I, Myers B, Minnis AM, Bonner CP, Ndirangu JW. Outcomes of substance use and sexual power among adolescent girls and young women in Cape Town: Implications for structural and cultural differences. Glob Public Health. 2024 Jan;19(1):2340500. doi: 10.1080/17441692.2024.2340500. Epub 2024 Apr 16. PMID 38628080
- [Derived] Singer SE, Wechsberg WM, Kline T, Browne FA, Howard BN, Carney T, Myers B, Bonner CP, Chin-Quee D. Binge drinking and condom negotiation behaviours among adolescent girls and young women living in Cape Town, South Africa: sexual control and perceived personal power. BMC Public Health. 2023 Nov 18;23(1):2282. doi: 10.1186/s12889-023-17188-0. PMID 37980472
- See also: The Young Women's Health CoOp in Cape Town, South Africa: Study protocol for a cluster-randomised trial for adolescent women at risk for HIV — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6042235/